CLINICAL TRIAL: NCT04393155
Title: Understanding Immunology and Patient Outcomes of COVID-19: A 1-Year Longitudinal Follow-up Study of Hospitalized Patients
Brief Title: COVID Cohort Study
Status: Terminated | Type: Observational
Why Stopped: Grant application to fund this work was not funded. We won't be posting data for this study.
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Professor of Medicine, University of Vermont
Other Study IDs: 16-540
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; Acute Respiratory Failure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19+: Hospitalized patients with acute respiratory failure (new oxygen requirement) due to COVID-19
  Interventions: Other: COVID-19+ observational

INTERVENTIONS:
Other: COVID-19+ observational — This is observational -- there is no intervention

SUMMARY:
The novel SARS-CoV-2 virus has quickly spread worldwide, with substantial morbidity and mortality. There is very limited understanding of the short- and longer-term inflammatory/immunological and clinical course. However, the investigators expect survivors from severe COVID-19 to experience persistent functional impairments, as demonstrated in prior studies of patients with acute respiratory distress syndrome (ARDS) and other acute viral illnesses. Notably, however, few studies have ever investigated the biologic mechanisms underlying these functional impairments. Understanding these features of COVID-19 will improve the ability to design acute therapies and recovery-focused interventions. To address these knowledge gaps, the investigators propose a two-center, 225 patient longitudinal prospective cohort study of hospitalized COVID-19 patients with acute respiratory failure. Researchers will perform an in-depth evaluation of inflammatory/immunological biomarkers, and physical, pulmonary, and neuropsychological clinical outcomes during hospitalization, and over 3-, 6-, and 12-month follow-up.

DETAILED DESCRIPTION:
The novel coronavirus (SARS-CoV-2) and associated COVID-19 illness has quickly spread worldwide, with substantial morbidity and mortality. Early data suggest that most patients with severe COVID-19 (i.e., experiencing acute respiratory failure (ARF) in an intensive care unit) may have cytokine release syndrome and other major effects on the innate and adaptive immune systems. However, there is limited understanding of both the inflammatory/immunological and the clinical course of COVID-19, with no robust data published beyond hospital discharge. Based on prior literature from acute viral illnesses, such as Ebola and Severe Acute Respiratory Syndrome (SARS), persistent functional impairments in COVID-19 survivors is expected. Despite the importance of these issues, very few studies have ever investigated the biological mechanisms underlying persistent functional impairments after ARF. Hence, understanding the short- and longer-term biological and clinical outcomes of patients with COVID-19, and investigating associations between inflammation and clinical outcomes is important to design acute therapies and recovery-focused interventions.

To address critical gaps in knowledge, the investigators propose a 2-center longitudinal cohort study of hospitalized COVID-19 patients via an Administrative Supplement to our existing grant (R01HL132887, MPIs Stapleton and Needham). Investigators will study COVID-19 patients with ARF who have either severe disease (requiring mechanical ventilation, non-invasive ventilation, or high flow nasal cannula oxygen support) or non-severe disease (new or increased supplemental oxygen requirement, without meeting severe criteria). Researchers will perform an in-depth evaluation of inflammatory/immunological, physical, pulmonary, and neuropsychological status during hospitalization, and over 3, 6, and 12-month follow-up. Feasibility for accomplishing this prospective study is demonstrated by 1) a successful existing collaboration between the University of Vermont (UVM) and Johns Hopkins University (JHU), supported by multiple NIH grants, and 2) the current and projected COVID-19 census at both hospital systems. The investigators have the existing infrastructure, expertise, and personnel to enroll 225 patients with COVID-19, and longitudinally follow survivors for 12 months, to investigate short-term and longer-term inflammatory/immunologic and clinical outcomes during this pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) at the time of consent
2. Positive COVID-19 test result or highly suspicious for COVID-19 infection and have a test pending
3. Acute Respiratory Failure (new requirement for supplemental oxygen or acute increase in required supplemental oxygen)

Exclusion Criteria:

1. Expected death or withdrawal of life-sustaining treatments within 3 days
2. Unable to walk ≥150 feet prior to COVID-19 (due to 6-minute walk test being primary outcome for in-person testing)
3. Hemoglobin ≤7.0 at the time of consent
4. Pre-existing cognitive/language impairment prohibiting clinical outcomes assessment
5. Prior lung resection (due to spirometry as part of in-person outcome assessment)
6. Unable to provide consent and no legally authorized representative (LAR) identified or reached by phone
7. Pregnant
8. Incarcerated
9. Homelessness
10. Physician declines patient enrollment (attending physician or study physician)
11. Patient or LAR do not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients hospitalized at participating medical centers who have a positive test result for COVID-19. These patients are expected to have a greater acuity of illness and burden of disease based on the fact that they require inpatient care. Enrolling hospitalized patients ensures a greater opportunity to collect serial biological specimens over the course of the illness due to proximity of the patient to medical and research staff and UVM laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Six minute walk distance (6MWD) | 3 months after hospital admission
  Exercise capacity

SECONDARY OUTCOMES:
Six minute walk distance (6MWD) | 6 months, 12 months after hospital admission
  Exercise capacity
Hospital Anxiety and Depression Scale (HADS) | 3 months, 6 months, 12 months after hospital admission
  Symptoms of anxiety and depression. Both anxiety and depression subscales are scored from 0-21, with higher scores indicating more symptoms.
EuroQol Group standardized measure of health status (EQ-5D-5L) | 3 months, 6 months, 12 months after hospital admission
  Health-related quality of life. The EQ-5D-5L is scored from 0-100, with a higher score indicating better health status.
MoCA-BLIND | 3 months, 6 months, 12 months after hospital admission
  Mental and Cognitive Functioning. The MoCA-BLIND is scored from 1-22, with higher scores indicating better cognitive function.
Health Care Utilization Survey (HUS) | 3 months, 6 months, 12 months after hospital admission
  Health Care Utilization
Death | 3 months, 6 months, 12 months after hospital admission
  Mortality
Forced vital capacity (FVC) | 3 months, 6 months, 12 months after hospital admission
  The maximum volume of gas expired when the patient exhales as forcefully and rapidly as possible after a maximal inspiration. Obtained by spirometry.
Forced expiratory volume in 1 second (FEV1) | 3 months, 6 months, 12 months after hospital admission
  Measure of the volume expired over the first second of an FVC maneuver. Obtained by spirometry
4-meter timed walk | 3 months, 6 months, 12 months after hospital admission
  Gait speed
Peripheral blood mononuclear cell type: CD4+ T cells (#cells/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Measured by cell staining and flow cytometry. PBMC differentiation/ activation/exhaustion status will be determined by multicolor flow cytometry staining with human monoclonal antibodies.
Peripheral blood mononuclear cell type: CD8+ T cells (#cells/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Measured by cell staining and flow cytometry. PBMC differentiation/ activation/exhaustion status will be determined by multicolor flow cytometry staining with human monoclonal antibodies.
Peripheral blood mononuclear cell type: B cells (#cells/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Measured by cell staining and flow cytometry. PBMC differentiation/ activation/exhaustion status will be determined by multicolor flow cytometry staining with human monoclonal antibodies.
Peripheral blood mononuclear cell type: NK cells (#cells/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Measured by cell staining and flow cytometry. PBMC differentiation/ activation/exhaustion status will be determined by multicolor flow cytometry staining with human monoclonal antibodies.
Peripheral blood mononuclear cell type: monocytes (#cells/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Measured by cell staining and flow cytometry. PBMC differentiation/ activation/exhaustion status will be determined by multicolor flow cytometry staining with human monoclonal antibodies.
Circulating markers of inflammation: C-Reactive Protein (CRP) (mg/l) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Interleukin 6 (IL-6) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Interleukin 8 (IL-8) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Interferon gamma (IFNg) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Interferon alpha (IFNa) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Tumor necrosis factor alpha (TNFa) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.
Circulating markers of inflammation: Interleukin 1 beta (IL-1b) (pg/ml) | study days 1, 3, and 7; then 3 months, 6 months, 12 months after hospital admission
  Biomarkers measured from plasma will be assayed using Luminex-based multiplex immunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided